# **Cover Page for ClinicalTrials.gov**

## Official Study Title:

Evaluation of a Cultural Dexterity Training Program for Surgeons: The PACTS Trial

### **NCT Number:**

NCT03576495

#### **Document:**

Statistical Analysis Plan

### **Document Date:**

June 6, 2017

PACTS ANALYSIS PLAN: The multi-year cluster-randomized study design will enable us to examine differences between and within the Early Intervention and Control/Delayed PACTS training groups across three unique time points (Year 2 pre-intervention, Year 2 post-intervention and Year 3 post-intervention). Details of statistical measures/methods and power calculations appear below.

Within-group differences (repeated measures). Repeated measure differences on dichotomous outcomes will be examined using Chi-square and Fisher's exact tests, as well as unadjusted logistic regression models controlling for resident-specific demographic factors (e.g. age, IAT, post-graduate year, and sex). Differences in ordinal outcomes (e.g. three- or

| Table 7. Sample Size Calculations | | | |
|---|---|---|---|
| Example | Proportional | Expected Minimum | Minimum Detectable Difference |
| Measure | Difference to be | Number of | (80% power and α=0.05) |
| | Measured | Participants Per | |
| | | Group | |
| Sample size/power calculations for repeated measures | | | |
| Within group | Pre-vs. Post-test | Pre-intervention: 160 | Pre-intervention: 50.0% |
| resident | proportion achieving | Post-intervention: | Post-intervention: 61.0% |
| knowledge/ | "Adequate" vs. "sub- | 160 | Thus, we expect to be able to detect a |
| skills/attitudes | optimal" dichotomized | (Repeated Measures) | proportional absolute difference of |
| | assessments | | 11% for within-group assessments. |
| | Sample size/power calculations for independent measures. | | |
| Between | Post-test proportion in | Early Group: 159 | Change from 50% to 65.5% |
| group resident | Early Group vs. | Delayed Group: 159 | Assuming remains at 50% with no |
| knowledge/ | Delayed Group | (Independent | change from baseline assessment. |
| Skills/attitudes | achieving "adequate" | Measures) | Thus, we would be able to detect a |
| | vs. "sub-optimal" | | 15% relative proportional difference |
| | dichotomized | | between groups associated with |
| | assessments | | exposure to PACTS training. |
| | Patient-reported within and between-group differences | | |
| Patient- | Pre-vs. Post-test | Pre-intervention: 361 | Proportion of Patients with scores |
| reported | proportion of patients | Post-intervention: | Pre-intervention: 63.0% |
| outcomes | reporting pain- | 361 | Post-intervention: 73.0% |
| | satisfaction scores in | (Independent | Thus, we expect to be able to detect |
| | the uppermost | Measures) | an absolute proportional difference of |
| | standardized quintile | | 10%. |
| Sample size/power calculation for NSQIP outcomes | | | |
| Readmissions | Pre- vs. Post-test | Pre-Intervention:377 | Proportion of Patients readmitted |
| | proportion of patients | Post-intervention:377 | Pre-intervention: 23% |
| | readmitted | | Post-intervention:15% |

five-point Likert scale reporting or ordered category scores) between pre- and post-intervention testing will be examined using Chi-square tests, unadjusted ordered logistic regression, and ordered logistic regression adjusted for resident- and program-specific factors. Table 7 depicts our sample size/power calculations, according to which we will be able to detect an 11% absolute difference in the proportion achieving "adequate" vs. "sub-optimal" dichotomized assessments before and after PACTS training. This accounts for an up to 20% sample loss from the expected 200 enrolled residents per group.

Table 7 Sample Size Calculations

**Between-group differences (independent measures).** Pre- vs. post- differences in both self-reported and observer-assessed ordinal outcomes between the Early and Delayed Intervention groups will be assessed at the end of the first training period using Chi-square tests and unadjusted ordered logistic regression, as well as ordered logistic regression models controlling for resident- and program-specific factors. Previous work demonstrated that exposure to training similar to PACTS was associated with a 20-25% increase in the proportion of trainees achieving "adequate" scores on an OSCE-based assessment. Based on the number of residents in each arm (n=200), we anticipate that we will be able to detect a much smaller between-group difference even with up to 20% sample attrition over time (Table 7).

*Pre- and post-intervention patient-reported satisfaction and NSQIP outcomes.* Management of pain will be assessed using elements of the Pain Treatment Satisfaction Scale (PTSS). Previous work by Gupta et al suggests that, on average, 63% of patients provided assessments of pain control satisfaction in the upper quintile of a standardized 10-point satisfaction scale. Subsequent to the intervention, it is estimated that 73% of patients treated by PACTS-trained residents will report satisfaction in the uppermost PTSS quintile. We expect an 8% decrease in readmissions, from 23% to 15% post-intervention. Pre-post intervention differences in patient-reported satisfaction and NSQIP outcomes will be assessed using Chi-square, Fisher's exact tests, or t-tests as appropriate, and ordinal scale differences will be assessed using Chi-Square tests and ordered logistic regression, both without adjustment and controlled for patient-, clinician-, and facility-level factors. It is important to note that the patient groups represent independent samples, and these pre- and post-intervention measures are independent measures, not repeated measures (Table 8). To achieve this, we will recruit 100 patients per site for each data collection phase. Thus, we will collect 300 patients per site over the entire study (2,400 total), giving ample power for both patient and clinical outcomes.